CLINICAL TRIAL: NCT00366925
Title: Randomized Controlled Multicenter Investigation to Compare the Efficacy and Safety of Adacolumn® Granulocytes, Monocytes/Macrophage Apheresis Device, 5 Versus 10 Treatments, in Patients With Active Ulcerative Colitis
Brief Title: CESA 5.10 Investigation to Compare the Efficacy and Safety of the Adacolumn® Apheresis Device in Patients With Active Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Frankfurt Research Institute GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Ada-UC-05-102
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Device: Adacolumn®

SUMMARY:
The purpose of this study is to compare the safety and efficacy of 5 Adacolumn® treatments over 5 weeks to 10 treatments (two Adacolumn® apheresis treatments during the first 2 weeks, followed by 6 weeks with one Adacolumn® apheresis treatment) in patients with active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old
2. Active ulcerative colitis documented by clinical symptoms, endoscopic findings and histology (in patient history)
3. Moderate to severe active ulcerative colitis at baseline evaluation, defined as follows:

   * Clinical activity idex (CAI) score > 6; and
   * Stool frequency score of 2 or 3
4. Colonic involvement with ulcerative colitis beyond 15 cm of the anal verge
5. Ulcerative colitis for at least 3 months
6. Adequate peripheral venous access to allow for completion of the apheresis treatments, as demonstrated by the ability to successfully undergo a brief venous access procedure
7. Receiving one or more of the following medical therapies:

   * Sulfasalazine, mesalamine and other 5-aminosalicylic acid (5-ASA) agents for 4 weeks or more with a stable dose for the last 2 weeks
   * A maximum of 20 mg per day of prednisone with a stable dose for the last 2 weeks, or
   * 6-mercaptopurine or azathioprine for 12 weeks or more with a stable dose for the last 4 weeks; OR

   Have not received the above medical therapies due to intolerance or demonstrated non-response for the time periods specified below:
   * Sulfasalazine, mesalamine and other 5-ASA agents for 2 weeks
   * Prednisone for 2 weeks, or
   * 6-mercaptopurine or azathioprine for 4 weeks
8. For female subjects of child-bearing potential, a negative pregnancy test and agreement to use an effective contraceptive method or abstain from sexual intercourse during the course of the clinical investigation
9. Agree to participate in the required follow-up visits
10. Able to complete the diary
11. Signed written informed consent document

Exclusion Criteria:

1. Febrile (> 38ºC)
2. Evidence of toxic megacolon
3. Anticipated need for surgery within 12 weeks
4. Known obstructive diseases of the gastrointestinal system
5. Proctocolectomy, total colectomy, ileostomy, stoma or ileal pouch-anal anastomosis
6. A history of allergic reaction to heparin or heparin-induced thrombocytopenia
7. A history of hypersensitivity reaction associated with an apheresis procedure or intolerance of apheresis procedures
8. Requires a central venous access catheter for the apheresis treatments
9. Known infection with enteric pathogens, pathogenic ova or parasites, or a positive assay for C. difficile toxin
10. Hypotension (systolic blood pressure < 90 mmHg and/or diastolic blood pressure < 65 mmHg) at screening visit only
11. Uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 120 mmHg) despite medical therapy at screening visit only
12. A history of myocardial infarction or unstable angina within the past 6 months
13. A history of coronary artery bypass grafting surgery or angioplasty within the past 6 months
14. A history of physical findings compatible with a cerebrovascular accident
15. Congestive heart failure (New York Heart Association Class III or IV)
16. Prosthetic heart valve, pacemaker or other permanent implant
17. Severe cardiovascular or peripheral vascular disease
18. Liver disease defined as levels of SGOT [AST], SGPT [ALT] or alkaline phosphatase > 2.5x the upper limit of the normal range for the laboratory performing test
19. History of cirrhosis
20. Renal insufficiency, defined as serum creatinine > 150% of the upper limit of the normal range for the laboratory performing the test
21. Insulin-dependent type I or type II diabetes. (Patients receiving oral antidiabetic treatment can be included.)
22. Known bleeding disorder (PT or PTT > 1.5x the upper limit of the normal range for the laboratory performing the test), or concomitant anticoagulant therapy for purposes other than apheresis treatment
23. Prior history suggestive of a hypercoagulable disorder, including 1 or more episodes of pulmonary embolism or deep vein thrombosis
24. Known infection with hepatitis B or C, or HIV
25. Abnormal hematology parameters defined as severe anemia with hemoglobin < 8.5 g/dL, white blood cell count of < 3,500/ul and a granulocyte count < 2,000/μl
26. Fibrinogen level > 700 mg/dL
27. Major surgery within the past 6 weeks
28. Infection:

    * Active infections less than 4 weeks from successful completion of antibiotic treatment for routine bacterial infection
    * Febrile viral infection within 4 weeks of entry into the clinical investigation
    * Less than 12 weeks from conclusion of therapy for systemic fungal infections
29. Malignancy within the past 2 years other than surgically cured skin carcinoma or cervical dysplasia (CIN I-II)
30. History of dysplasia or carcinoma of the colon
31. Current drug or alcohol abuse
32. Pregnant, lactating or planning to become pregnant during the course of the clinical investigation
33. Used within the last 30 days, an investigational drug, biologic or device or 5 half lives, if known, for any investigational drug or biologic
34. Received cyclosporine or tacrolimus within the last 4 weeks
35. Received infliximab within the last 8 weeks
36. Received oral budesonide within the last 2 weeks
37. Used topical therapy for ulcerative colitis within the last 2 weeks
38. Previously received Adacolumn® treatments

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Dignass, Prof. Dr. med., Principal Investigator — Markus-Krankenhaus, Frankfurt am Main
Locations (1):
- Markus-Krankenhaus, Frankfurt am Main, Hesse, Germany